CLINICAL TRIAL: NCT06242600
Title: A Prospective Single-center Randomized Pilot Study to Evaluate the Safety and Performance of the Novel CytaCoat LIP Foley Catheter When Compared to an Uncoated Foley Catheter
Brief Title: Evaluation of Safety and Performance of the CytaCoat Lubricious Infection Prevention (LIP) Foley Catheter
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CytaCoat AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIV-23-03-042616; CYTA-FOL-1 (Other: CytaCoat)
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Safety of the CytaCoat LIP Foley Catheter; Tolerability of the CytaCoat LIP Foley Catheter

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to CytaCoat LIP Foley catheter / uncoated silicone Foley catheter (15 patients in each arm).
Who Masked: Outcomes Assessor
Masking Description: The healthcare practitioner placing the catheter will know the allocation (whether it is a CytaCoat LIP Foley catheter or the comparator) but the participant will not know which catheter they have received.
  The healthcare practitioner removing the catheter will not know the allocation. Urine samples that are analysed will not state which arm the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CytaCoat LIP Foley catheter (Experimental): CytaCoat LIP Foley catheters will be randomized 1:1 (15 patients in each arm), to patients in need of catheterization for up to 24 hrs.
  Interventions: Device: Drainage of the bladder by indwelling Foley catheter
- Uncoated silicone Foley catheter (Other): Uncoated silicone Foley catheter will be randomized 1:1 (15 patients in each arm), to patients in need of catheterization for up to 24 hrs.
  Interventions: Device: Drainage of the bladder by indwelling Foley catheter

INTERVENTIONS:
Device: Drainage of the bladder by indwelling Foley catheter — Drainage of the bladder by transurethral catheterization with an indwelling Foley catheter of patients undergoing a TUR-B procedure and in need of a Foley catheter for up to 24 hrs.
  Other Names: CytaCoat LIP Foley catheter

SUMMARY:
The goal of this pilot safety and tolerability study is to determine whether the novel CytaCoat LIP (Lubricious Infection Prevention) Foley catheter is safe to use in patients during short term use.

The primary objective of this study is to determine the safety and tolerability for the medical device CytaCoat LIP Foley catheter in patients undergoing Transurethral Resection of the Bladder (TUR-B) surgery. Safety will be assessed by evaluation of adverse events.

The secondary objective is to assess the overall performance by evaluating if there were any Foley catheter handling problems experienced by the healthcare personnel with the use of the CytaCoat LIP Foley catheter.

Exploratory objectives are to assess bacterial culture of urine samples taken before and after catheterization and to assess pain, irritation and discomfort measured by asking patients about their experience using the catheter using a questionnaire.

Participants will be catheterized with either a CytaCoat Foley catheter or an uncoated silicone catheter, for a maximum of 24 hrs. After removal of the catheter, participants will be asked to assess if they experienced any pain, irritation and discomfort measured with the Numerical Rating Scale (NRS) (0-10). A similar assessment will be performed 7-10 days after removal of the catheter. In addition, the healthcare personnel will be asked to assess the functionality of the coated catheter with the NRS scale (0-10), using a questionnaire. Urine samples will be taken before and after catheterization and evaluated through quantification.

ELIGIBILITY:
Inclusion Criteria:

* Will be undergoing a TUR-B procedure.
* Able to give informed consent by signing and dating the written informed consent document acknowledging their desire to participate in the study.
* Adults, age 18 to 84 years.
* Require insertion of a size 12, 14, 16, 18 or 20 French Foley catheter after TUR-B surgery.
* Be able to understand and comply with the information given in the Patient Consent Form.

Exclusion Criteria:

* Vulnerable subjects such as children, pregnant or breastfeeding women, or potentially immune-compromised subjects.
* Unable to provide informed consent.
* Has a known bacteriuria or a current urinary tract infection.
* Has a known bloodstream infection or an infection that requires prolonged antibiotic therapy.
* Has an ongoing antibiotic therapy.
* Cannot accommodate a size 12, 14, 16, 18 or 20 Fr Foley catheter or requires a Thiemann tip Foley catheter.
* Previous enrolment in the present study.
* Simultaneous participation in another clinical study that may impact the primary endpoint.
* Severe non-compliance to protocol as judged by the PI.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Assessment of incidence of adverse events and serious adverse events (safety and tolerability) of the CytaCoat LIP Foley catheter | 1 - 10 days
  Adverse events (AEs) and serious adverse events (SAEs) will be assessed, which are further divided into adverse device effects (ADEs) and serious ADEs (SADEs).

SECONDARY OUTCOMES:
Assessment of the overall performance of the CytaCoat LIP Foley catheter | 1 - 10 days
  The functionality of the coated catheter will be assessed by a responsible nurse/physician with the NRS scale (0-10) using questionnaires.

OTHER OUTCOMES:
Exploratory assessment of bacterial culture of urine samples | 1 - 48 hours
  Assessment by quantitative bacterial culture of urine samples obtained from patients when first included in the study and subsequently after clamping the catheter for 30 minutes prior to extirpation of the catheter.
Exploratory assessment of patient user experience of the CytaCoat LIP Foley catheter | 1 - 10 days
  Assessment immediately after removal of the catheter of pain, irritation and discomfort measured with the NRS scale (0-10) using a questionnaire asking patients about their experience using the catheter.
  Assessment 7-10 days after removal of the catheter of pain, irritation and discomfort measured with the NRS scale (0-10) using a questionnaire asking patients about their experience using the catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Andreasson, MD, Principal Investigator — Sahlgrenska University Hospital, Department of Urology
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No